CLINICAL TRIAL: NCT04998110
Title: Pilot Randomized Controlled Trial of Integrated Palliative Care With Nephrology Care
Brief Title: Integrated Palliative Care With Nephrology Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-00507; K23DK125840-02 (NIH)
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: CKD

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Care Intervention (Experimental): The supportive care intervention arm will receive their usual ambulatory longitudinal nephrology care integrated with ambulatory supportive care through monthly supportive care visits over six months.
  Interventions: Other: Ambulatory Supportive Care
- Usual Care Control (No Intervention): The usual care control arm will be seen at the discretion of their nephrologist, or receive their usual dialysis if on dialysis.

INTERVENTIONS:
Other: Ambulatory Supportive Care — Ambulatory supportive care visits monthly for six months - a monthly visit with an ambulatory palliative care provider educated in kidney disease
  Arms: Supportive Care Intervention

SUMMARY:
This study is a pilot randomized controlled trial testing the effectiveness of integrated ambulatory supportive care visits with standard nephrology outpatient visits for six months in patients with advanced CKD. The study team hypothesizes that patients in the integrated care arm will trend towards improved symptom burden, improved quality of life scores and more engagement in advance care planning.

Primary objectives: To test the impact of integrated ambulatory supportive care in nephrology care on symptom burden. Secondary: To test the impact of integrated ambulatory supportive care on quality of life and engagement in advance care planning and to demonstrate study feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Documented diagnosis of Chronic Kidney Disease stage IV or V
3. Speaks Spanish or English fluently
4. Provision of signed and dated informed consent form
5. Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study.

Exclusion Criteria:

1. Exposure to supportive/palliative care in the last six months either inpatient or outpatient.
2. Presence of a condition(s) or diagnosis, either physical or psychological, or physical exam finding that precludes participation, for example not being able to cognitively understand the questions or to provide informed consent.
3. Pregnant women.
4. Not fluent in either English or Spanish
5. Any urgent supportive/palliative care needs identified on screening interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Month 12
  This will be reported as the percentage of participants who provide informed consent.
Number of Participants who Maintain Participation in the Study (Retention) | Month 12
  Reported as percentage of participants who signed informed consent, who completed the study.
Average number of clinical visits attended per participant (Retention) | Month 12
Ability to Collect Planned Data | Month 12
  This will be reported as the percent of completed data surveys

SECONDARY OUTCOMES:
Change in Kidney Disease Quality of Life (KDQOL-36) Score | Baseline, Month 6
  The KDQOL is a 36-item quality of life survey that includes five domains: Physical Component Summary (PCS), a Mental Component Summary (MCS), Burden of Kidney Disease Score, Symptoms and Problems of Kidney Disease Score, and Effect of Kidney Disease Score. All scores are on a scale of 0-100, with higher scores representing better quality of life.
Engagement in Advance Care Planning | Baseline, Month 6
  Advance care planning will be measured by total number of advance care planning conversations held.
Change in Integrated Palliative Outcome Score-Renal (IPOS-Renal) Score | Baseline, Month 6
  The scoring will include 11 questions on the degree of impact kidney-specific symptoms have had on patients over the past week, plus additional items on concerns beyond symptoms, such as information needs, practical issues, and family anxiety. This includes one question that has 15 sub-questions asking about specific physical symptoms. All scores are on a scale of 0-90, with lower scores representing less problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Scherer, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYC Health + Hospitals / Bellevue, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Jennifer.scherer@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Scherer JS, Wu W, Lyu C, Goldfeld KS, Brody AA, Chodosh J, Charytan D. A pilot randomized controlled study of integrated kidney palliative care and chronic kidney disease care implemented in a safety-net hospital: Protocol for a pilot study of feasibility of a randomized controlled trial. Contemp Clin Trials Commun. 2025 Feb 3;44:101439. doi: 10.1016/j.conctc.2025.101439. eCollection 2025 Apr. PMID 40008278

DOCUMENTS (1):
  • Informed Consent Form (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT04998110/ICF_000.pdf